CLINICAL TRIAL: NCT06693323
Title: Single-Center Evaluation of the Clinical and Radiological Benefit of AHCC® in Combination with Standard of Care Treatment for HPV-Positive Patients with Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Single-Center Eval of Clinical & Radiological Benefit AHCC in Combo W/ SOC Tx for HPV+ Pts W/ HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Rupali Nabar, Associate Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5821; UCI 21-173 (Other: UCI CFCCC)
Record Dates: First submitted 2024-11-13; First posted 2024-11-18 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: HNSCC; Head and Neck Squamous Cell Carcinoma
Keywords: HNSCC; Head and Neck Squamous Cell Carcinoma; AHCC; HPV-Positive HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AHCC (Experimental): Oral Drug
  Interventions: Drug: AHCC®capsules

INTERVENTIONS:
Drug: AHCC®capsules — Given PO

SUMMARY:
This is a phase 2, single-arm, open-label clinical trial determining safety and tolerability of AHCC in subjects with HPV-positive patients with Head and Neck Squamous Cell Carcinoma. These are subjects who have undergone surgery or will be undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 79 years of age.
* Has a diagnosis of pathologically or cytologically proven HPV positive HNSCC.
* For patients who have undergone surgery, they must be registered at least 4 weeks after surgery.
* For patients that have completed surgery, has a high risk disease defined as:

  1. Positive Margins and/or Extra Nodal Extension (ENE)
  2. Positive margins are defined as malignancy at or within 1 mm of the margin. High grade dysplasia (i.e., carcinoma in situ) at the margin is also considered positive
  3. ENE may be either gross or microscopic
* No evidence of distant disease based on baseline imaging done within 28 days prior to registration. Patient may be any T or N stage, but must be M0
* Has an ECOG Performance Status 0-1.
* Has the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible.
* All females of childbearing potential must have a blood test or urine study within 14 days prior to registration negative for pregnancy.

  1. A female of childbearing potential is defined as any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets any of the following criteria: has achieved menarche at some point, has not undergone a hysterectomy or bilateral oophorectomy, or has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* Women of childbearing potential and sexually active males must not conceive or father children by using accepted and effective method(s) of contraception or by abstaining from sexual intercourse while on study treatment, and continue for 120 days after the last dose of study treatment. Accepted and effective methods are described in Appendix 4
* Has adequate organ and marrow function as defined below, based on clinical laboratory assessments obtained ≤ 28 days prior to registration:

  1. Absolute neutrophil count (ANC) ≥ 1,500/μL
  2. Platelets ≥ 100,000/μL
  3. Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN)
  4. AST or /ALT ≤ 3.0 × institutional ULN
  5. Creatinine clearance > 30 mL/min using the Cockcroft-Gault formula

Exclusion Criteria:

* Patient must not be pregnant or breast-feeding due to the unknown potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used.
* Current active infection that requires systemic treatment at time of registration.
* History of solid organ transplant or stem cell transplant.
* Currently taking immunosuppressive medication within 7 days prior to registration, EXCEPT for the following:

  1. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection)
  2. systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent
  3. steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* New York Heart Association Class III or IV heart failure. Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification.
* Received a live vaccine within 30 days prior to the first dose of study drug.

  1. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), or typhoid fever.
  2. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
  3. COVID-19 (SARS-CoV-2) vaccines (mRNA or other) are allowed.
* Known history of Hepatitis B (defined as HBsAg reactive) or known active Hepatitis C virus (defined as positive for HCV RNA on a qualitative test).
* History of HIV with or without antiviral treatment having

  1. detectable viral loads within 6 months, or
  2. history of Kaposi sarcoma and/or Multicentric Castleman Disease.
* Active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* Known allergy to mushrooms, mushroom products, or any components of the study formulation.
* Known psychiatric or substance abuse disorder that would interfere with the participant's ability to complete study assessments or to adhere to protocol requirements.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) of Patients receiving AHCC and concurrent standard of care treatment regimens | 60 months
  To evaluate the overall survival of patients with HPV-positive Head and Heck squamous cell carcinoma

SECONDARY OUTCOMES:
Difference in Tumor Response of patients receiving concurrent therapy with chemoradiation plus AHCC over SoC treatment and in the long term follow up period compared to historical data. | 5 years
  Tumor response will be assessed by RECIST 1.1 consist of a standardize set of imaging procedures with results graded using the American Joint Committee on Cancer TNM staging system version 8.
Percentage of Adverse Events | Up to 24 cycles
  To evaluate safety and tolerability of AHCC in HPV+ patients with HSNCC receiving concurrent SoC treatment regiments by estimating proportion of adverse events for the following patients who experience at least one of the following:
  1. Neutropenia adverse event at a grade of 3 or above
  2. Neutropenia adverse event
  3. Renal impairment adverse event
  4. Hepatic dysfunction adverse event
  5. Neuropathy event
  6. Ototoxicity adverse event

OTHER OUTCOMES:
Change in Quality of Life (QoL) score | At the end of Cycle 6 (each cycle is 28 days)
  QoL score measurement will be defined as the change from baseline to Cycle 6
Changes in HPV DNA in blood samples from HPV+ patients with HNSCC | Up to 5 years
  Evaluate whether changes in HPV DNA in blood samples from HPV+ patients with HNSCC have predictive value as a marker of tumor response or recurrence in HPV+ patients that have received SoC treatment regimens

CONTACTS AND LOCATIONS:
Overall Officials: Rupali Nabar, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, University of California, Irvine, Orange, California, United States